CLINICAL TRIAL: NCT00510341
Title: Asthma Management Support Training in Pediatrics
Brief Title: Evaluating the Collaborative Management in Pediatrics (CMP) Training Program Among Pediatric Resident Doctors and Their Patients With Asthma or Obesity
Acronym: CMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 405; R21HL080067-01 (NIH)
Record Dates: First submitted 2007-07-31; First posted 2007-08-02 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Education; Asthma; Obesity
Keywords: Behavior Change Counseling; Motivational Interviewing; Chronic Care Model; Communication; Residency Training; Skill Assessment
MeSH Terms: conditions — Asthma; Obesity; Communication | interventions — Cytidine Monophosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): CMP program
  Interventions: Behavioral: Collaborative Management in Pediatrics (CMP) Program
- 2 (No Intervention): Control group

INTERVENTIONS:
Behavioral: Collaborative Management in Pediatrics (CMP) Program — Pediatric residents will receive two 4.5 hour training sessions on the CMP Program.
  Arms: 1

SUMMARY:
Self-care behaviors are decisions and actions that people can take to improve their health or cope with a health problem. It is important for people with long-term illnesses to develop and maintain effective self-care behaviors. This study will evaluate the usefulness and practicality of the Collaborative Management in Pediatrics (CMP) program, which is a training program developed to encourage pediatric resident doctors to promote self-management of illness and behavior change among children with asthma or obesity and their families.

DETAILED DESCRIPTION:
Collaborative management health care involves strengthening and supporting self-care among people with long-term illnesses while assuring that effective medical, preventive, and health maintenance treatments occur. In collaborative management, it is important for patients, family members, and health care providers to understand each other's roles and responsibilities as they work toward a shared goal of improving the patient's health. Examples of self-care behaviors include reading books or other materials about relevant health care topics, exercising, following a low-fat diet, seeing a doctor on a regular basis, and making lifestyle changes. It is crucial that doctors, case managers, nurses, pharmacists, and other medical professionals understand the challenges that patients face when attempting to incorporate these self-care behaviors into their lives. Currently, there are few collaborative management programs that specifically address pediatric long-term illness and even fewer programs that identify doctors as the primary medical professional responsible for encouraging behavior change.

The CMP program will incorporate a collaborative management technique with a motivational interviewing approach. Motivational interviewing is a counseling style that attempts to increase awareness of the potential problems, causes, consequences experienced, and risks faced as a result of the behavior in question. The goal of the CMP program is to help pediatric resident doctors accomplish the following: assess patients' asthma and obesity status and related health behaviors; assess the child/family aspect of self-care; motivate parents and children to change asthma or obesity health behaviors; collaboratively set goals for asthma management by the family; and provide tailored follow-up to patients and their families. The purpose of this study is to evaluate the feasibility of the various components of the CMP program. Results from this study will be used to develop a larger clinical trial that will evaluate the effectiveness of the CMP program.

This pilot study will enroll 18 first-year pediatric resident doctors; each doctor will select five of their pediatric patients with asthma or obesity to participate in the study. Each resident doctor will be randomly assigned to take part in either the CMP program or a control group. All resident doctors will complete an Objective Structured Clinical Examination (OSCE), which will be used to assess their skills and ability in the areas of communication, clinical examination, medical procedures, prescribing medication, and interpretation of test results. Resident doctors participating in the CMP program will then receive CMP training. Three weeks following the initial OSCE, all resident doctors will perform a repeat OSCE, which will evaluate the effectiveness of the CMP training. One health care visit will then be conducted with each participating patient. During this visit, the resident doctor will conduct a collaborative management session emphasizing the family's central role in managing the child's health. Study researchers will conduct a 30-minute telephone interview with the child's parents at baseline, Week 6, following the heath care visit, and Month 3. Parent/child behaviors, attitudes related to asthma or obesity, management of their child's health, and satisfaction with care will be assessed during the telephone interviews. All residents will complete a repeat OSCE at Month 6 to assess any increase or decrease in skills.

ELIGIBILITY:
Inclusion Criteria for Pediatric Resident Doctors:

* Attends the University of Washington's pediatric residency program and has a continuity clinic at one of the three participating sites (Odessa Brown Children's Clinic, Pediatric Care Center, or Harborview's Children and Teens Clinic)

Inclusion Criteria for Child Participants:

* Diagnosed with either asthma or obesity and on the continuity panel of a participating resident doctor

Exclusion Criteria for Pediatric Resident Doctors:

* Previously participated in the project development of the CMP training

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2006-04; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Feasibility and acceptability of various components of the CMP program | Measured at the completion of the 1-year study

SECONDARY OUTCOMES:
Effect size of CMP training on resident skills and patient-centered outcomes | Measured at the completion of the 1-year study
Reliability of the OSCEs, which are used to assess resident skill | Measured at the completion of the 1-year study

CONTACTS AND LOCATIONS:
Overall Officials: Paula Lozano, MD, MPH, Principal Investigator — Child Heatlh Institute, University of Washington
Locations (3):
- United States (3):
  - Harborview's Children and Teens Clinic, Seattle, Washington
  - Pediatric Care Center, Seattle, Washington
  - Odessa Brown Children's Clinic, Seattle, Washington

REFERENCES:
- [Derived] Lozano P, McPhillips HA, Hartzler B, Robertson AS, Runkle C, Scholz KA, Stout JW, Kieckhefer GM. Randomized trial of teaching brief motivational interviewing to pediatric trainees to promote healthy behaviors in families. Arch Pediatr Adolesc Med. 2010 Jun;164(6):561-6. doi: 10.1001/archpediatrics.2010.86. PMID 20530307